CLINICAL TRIAL: NCT01708993
Title: A Randomized Phase II Study of Reolysin in Patients With Previously Treated Advanced or Metastatic, Non Small Cell Lung Cancer Receiving Standard Salvage Therapy.
Brief Title: Reolysin in Previously Treated Advanced/Metastatic, Non Small Cell Lung Cancer Receiving Standard Salvage Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I211
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; reolysin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: Pemetrexed and Reolysin (and safety run-in) (Active Comparator)
  Interventions: Drug: Pemetrexed and Reolysin (and safety run-in)
- Arm B: Pemetrexed (Active Comparator)
  Interventions: Drug: Pemetrexed
- Arm C: Docetaxel and Reolysin (and safety run-in) (Active Comparator)
  Interventions: Drug: Docetaxel and Reolysin
- Arm D: Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Pemetrexed and Reolysin (and safety run-in) — Pemetrexed: 500 mg/m², IV (10 min) - Day 1 every 3 weeks Reolysin: 4.5 x 10^10 TCID50 IV (1 hour) - Days 1-3, every 3 weeks
  Arms: Arm A: Pemetrexed and Reolysin (and safety run-in)
Drug: Pemetrexed — Pemetrexed: 500 mg/m² IV (10 min) - Day 1 every 3 weeks
  Arms: Arm B: Pemetrexed
Drug: Docetaxel and Reolysin — Docetaxel: 75 mg/m² IV (1 hour) - Day 1 every 3 weeks Reolysin: 4.5x10^10 TCID50 IV (1 hour) - Days 1-3, every 3 weeks
  Arms: Arm C: Docetaxel and Reolysin (and safety run-in)
Drug: Docetaxel — Docetaxel: 75 mg/m² IV (1 hour) - Day 1 every 3 weeks
  Arms: Arm D: Docetaxel

SUMMARY:
The purpose of this study is to find out if giving reolysin in combination with docetaxel or pemetrexed can offer better results than standard therapy with docetaxel or pemetrexed alone.

DETAILED DESCRIPTION:
Reolysin is a virus which has been shown to target and destroy cancer cells in laboratory tests. Reolysin has been studied in over 360 cancer patients to find safe doses that can be given and has also undergone testing in combination with docetaxel.

Docetaxel and pemetrexed have anticancer activity in certain cancers including lung and they have been approved by Health Canada for the treatment of patients with advanced or metastatic non-small cell lung cancer.

Researchers doing this study also want to evaluate the side effects of reolysin when given together with docetaxel or pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC). As treatment arm is assigned based on histology subtype, it must be feasible to subtype into squamous or other.
* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available for translational studies and must have provided informed consent for the release of the block as well as for blood samples for correlative studies.
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:

  * Chest X-ray ≥ 20 mm
  * CT/MRI scan (with slice thickness of < 5 mm) ≥ 10 mm --> longest diameter
  * Physical exam (using calipers) ≥ 10 mm
  * Lymph nodes by CT scan ≥ 15 mm --> measured in short axis All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative).
* Patients must have advanced and or metastatic disease, for which no curative therapy exists and for which systemic therapy is indicated.
* ECOG performance of 0 or 1.
* Age ≥ 18 years.

Surgery: Previous major surgery is permitted provided that it has been at least 14 days prior to patient randomization and that wound healing has occurred.

Chemotherapy: Patients must have received one regimen of palliative first line chemotherapy (must be platinum containing combination unless patient's age > 70 years) which may not have contained docetaxel. Patients who have had concurrent platinum based chemoradiotherapy for stage three disease and have relapsed within one year of treatment, or patients who have had platinum based adjuvant chemotherapy after complete surgical resection and have relapsed within one year of treatment, may be considered to have had one prior platinum containing regimen.

Prior paclitaxel is permissible. Patients who have had prior pemetrexed for first line therapy will be randomized to Treatment Arm C or D (docetaxel ± reolysin). Prior maintenance therapy with pemetrexed is not permitted. Prior adjuvant chemotherapy is permissible providing completed at least 1 year prior to relapse/recurrence of disease and the patient has received one regimen of palliative first line chemotherapy as described above.

Other Therapy: Patients may have received other therapies including immunotherapy, or with signal transduction inhibitors, including EGFR inhibitors.

Radiation: Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, non-myelosuppressive radiotherapy.

* Laboratory Requirements (must be done within 7 days prior to randomization)

  * Hematology:
  * Neutrophils ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Biochemistry:
  * Serum creatinine ≤ 1.5 x ULN (For patients enrolled to a pemetrexed arm, the creatinine clearance must also be >45 ml/min)
  * Total bilirubin ≤ 1.0 x ULN (unless elevated secondary to conditions such as Gilbert's disease)
  * ALT and AST ≤ 1.5 x ULN (≤ 3x ULN is permitted in the presence of known liver metastases)
  * Proteinuria <2g/24hrs (screen using spot testing; if ≥ grade 2 repeat with mid-stream urine; if still ≥ grade 2 then uring collection for 24 hours to confirm <2g/24hrs).
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumours curatively treated with no evidence of disease for > 3 years.
* Patients who are on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients with significant cardiac (including uncontrolled hypertension) or pulmonary disease, or active CNS disease or infection.
* Patients with a known hypersensitivity to the study drug(s) or their components.
* Patients with untreated brain metastases, untreated spinal cord compression or meningeal metastases are not eligible (CT scans are not required to rule this out unless there is a clinical suspicion of CNS disease). Patients with treated brain metastases who have radiologic evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to randomization).
* Patients who have neuropathy ≥ grade 2 (patients planned for docetaxel Arms C and D only).
* Women must be post-menopausal, surgically sterile or use two reliable forms of contraception while on study and for 6 months after discontinuing therapy. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to registration/randomization and must not be lactating. Men must be surgically sterile or use a barrier method of contraception.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 30 months
  Evaluation of the effect of reolysin in combination with standard salvage chemotherapy on the progression free survival of patients with advanced or metastatic NSCLC. Response and progression will be evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee

SECONDARY OUTCOMES:
Number of patients with adverse events | 30 months
  To determine the tolerability and toxicity of reolysin and standard salvage chemotherapy when given in combination.
Response rates | 30 months
  To investigate additional potential measures of efficacy including:
  * Progression rates at 3 months
  * Objective response rate
  * Overall survival (OS)
Explore potential molecular factors predictive of response | 30 months
  Exploration of potential molecular factors predictive of response by assessment of archival tumour tissue and serial blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Donald G Morris, Study Chair — Tom Baker Cancer Centre, Calgary Alberta Canada
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bradbury PA, Morris DG, Nicholas G, Tu D, Tehfe M, Goffin JR, Shepherd FA, Gregg RW, Rothenstein J, Lee C, Kuruvilla S, Keith BD, Torri V, Blais N, Hao D, Korpanty GJ, Goss G, Melosky BL, Mates M, Leighl N, Ayoub JP, Sederias J, Feilotter H, Seymour L, Laurie SA. Canadian Cancer Trials Group (CCTG) IND211: A randomized trial of pelareorep (Reolysin) in patients with previously treated advanced or metastatic non-small cell lung cancer receiving standard salvage therapy. Lung Cancer. 2018 Jun;120:142-148. doi: 10.1016/j.lungcan.2018.03.005. Epub 2018 Mar 9. PMID 29748010